CLINICAL TRIAL: NCT03366220
Title: Resuscitation With Plasma in Surgical and Trauma Patients With Septic Shock
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was halted early due to low patient accrual secondary to COVID-19 and significant heterogeneity in clinical manifestations of sepsis precluding enrollment.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Lillian Kao, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HSC-MS-17-0714
Record Dates: First submitted 2017-12-01; First posted 2017-12-08 (Actual); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Septic Shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- initial resuscitation with plasma (Experimental): Initial resuscitation with plasma will be 10 mL/kg (700 mL in a typical 70 kg adult). Traditional doses of plasma, when used to correct coagulopathy range from 10-15 mL/kg.23 The plasma will be administered at a rate of 2-3 mL/kg/hr (140-210 mL/hr in a typical 70 kg adult). A research physician will be at bedside to follow patient resuscitation. Plasma administration may be terminated before the entire dose is administered if patients show clinical improvement. After the initial dose of plasma has been given, subsequent resuscitation will follow usual care using balanced crystalloids.
  Interventions: Drug: Plasma
- initial resuscitation with balanced crystalloids (Active Comparator): Usual care using balanced crystalloids (Iso-Lyte or Plasma-Lyte) only will follow Surviving Sepsis Campaign guidelines. Controls will receive 30 mL/kg (2100 mL in a typical 70 kg adult) of crystalloids within the first 3 hours. Subsequent resuscitation with balanced crystalloids will be titrated to the endpoints of resuscitation.
  Interventions: Drug: Balanced crystalloids

INTERVENTIONS:
Drug: Plasma — Initial resuscitation with plasma will be 10 mL/kg (700 mL in a typical 70 kg adult). Traditional doses of plasma, when used to correct coagulopathy range from 10-15 mL/kg.23 The plasma will be administered at a rate of 2-3 mL/kg/hr (140-210 mL/hr in a typical 70 kg adult). A research physician will be at bedside to follow patient resuscitation. Plasma administration may be terminated before the entire dose is administered if patients show clinical improvement. After the initial dose of plasma has been given, subsequent resuscitation will follow usual care using balanced crystalloids.
  Arms: initial resuscitation with plasma
Drug: Balanced crystalloids — Usual care using balanced crystalloids (Iso-Lyte or Plasma-Lyte) only will follow Surviving Sepsis Campaign guidelines. Controls will receive 30 mL/kg (2100 mL in a typical 70 kg adult) of crystalloids within the first 3 hours. Subsequent resuscitation with balanced crystalloids will be titrated to the endpoints of resuscitation.
  Arms: initial resuscitation with balanced crystalloids

SUMMARY:
There is a knowledge gap regarding the optimal initial fluid to achieve effective resuscitation and improved outcomes in septic shock. The purpose of this study is to compare initial resuscitation with plasma to initial resuscitation with balanced crystalloids.

ELIGIBILITY:
Inclusion Criteria:

* Patients meeting the following criteria will be enrolled: Have a Sepsis Screening Score (SSS) ≥ 4 with a suspected source of infection (Table 1); and Written informed consent obtained
* Patients meeting any of the following criteria will be randomized: Hypotension with MAP < 65 mmHg; Lactic acid > 4 mmol/L; Altered mental status; and Decreased urine output of < 0.5 mL/kg in the past hour.

Exclusion Criteria:

* Pregnancy
* Prisoners
* Traumatic brain injury
* Evidence of ongoing hemorrhage, history of congenital bleeding disorders, therapeutic anticoagulation
* History of myocardial infarction or congestive heart failure
* History of acute cerebral vascular event
* Major burns (>20% total body surface area)
* History of adverse reactions to blood product transfusion
* Contraindications to blood transfusions (eg. Jehovah's Witness)
* Contraindications to central venous line and arterial line placement
* On intermittent hemodialysis
* Do-Not-Resuscitate or Comfort Care status
* Participation in another interventional study
* Pending transfer to another unit within the hospital that is not STICU or SIMU

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-26 (Actual); Primary Completion 2019-09-17 (Actual); Study Completion 2019-10-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shuyan Wei, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

REFERENCES:
- [Derived] Wei S, Kao LS, Wang HE, Chang R, Podbielski J, Holcomb JB, Wade CE. Protocol for a pilot randomized controlled trial comparing plasma with balanced crystalloid resuscitation in surgical and trauma patients with septic shock. Trauma Surg Acute Care Open. 2018 Sep 23;3(1):e000220. doi: 10.1136/tsaco-2018-000220. eCollection 2018. PMID 30271882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients with a sepsis screening score > or equal to 4 (which indicates potential sepsis) and with a suspected source of infection were enrolled, and they were later randomized if septic shock developed, per the protocol. Only 8 enrolled patients progressed to septic shock, and therefore only 8 participants were randomized and started the protocol.
Period: Overall Study
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.75 (9.81) | 58 (9.09) | 44.37 (9.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 0 | 3 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 2 | 5
  Black | 1 | 2 | 3
  Hispanic | 0 | 0 | 0
  Other | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Glycocalyx Breakdown as Assessed by Syndecan-1 Levels
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and at 24 hours
Population: Data was not collected at end of initial bolus of fluid administration (about 3 hours) and 24 hours for one participant in the initial resuscitation with balanced crystalloids arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
ng/mL
  0 hours | 260.87 (455.79) | 390.67 (169.66)
  2 hours | 294.03 (499.12) | 383.53 (122.26)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 278.22 (456.24) | 337.37 (220.03)
  12 hours | 291.28 (496.24) | 350.43 (196.62)
  24 hours: number analyzed (Participants) | 4 | 3
  24 hours | 241.16 (349.15) | 285.34 (45.10)

2. Primary Outcome: Glycocalyx Breakdown and Endothelial Leakage as Assessed by Soluble Thrombomodulin (sTM)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: Data was not collected at end of initial bolus of fluid administration (about 3 hours) and at 24 hours for one participant in the initial resuscitation with balanced crystalloids arm.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
ng/mL
  0 hours | 22.44 (14.94) | 21.29 (12.22)
  2 hours | 22.06 (17.19) | 21.50 (11.66)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 21.87 (15.88) | 23.38 (14.28)
  12 hours | 21.13 (12.59) | 22.10 (11.86)
  24 hours: number analyzed (Participants) | 4 | 3
  24 hours | 25.69 (21.02) | 24.43 (12.78)

3. Primary Outcome: Endothelial Leakage as Assessed by Soluble FMS-like Tyrosine Kinase-1 (sFLT-1)
Time Frame: 0, 2, end of initial bolus of fluid administration(about 3 hours), 12, and 24 hours
Population: Data was not collected for this outcome measure.
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Endothelial Leakage and Inflammation as Assessed by Vascular Endothelial Growth Factor (VEGF)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: In the plasma arm, sample levels were out of range and thus no value could be obtained for 3 participants at all time points.
  In the balanced crystalloids arm, sample levels were out of range and thus no value could be obtained for 3 participants at 0, 2, and 12 hours; for 2 at about 3 hours and at 24 hours; and for all 4 at 12 hours--in addition to those with sample levels out of range, there was 1 other participant for whom no data at all were collected at 3 hours and 24 hours.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours: number analyzed (Participants) | 1 | 1
  0 hours | 108.35 (0) | 61.6 (0)
  2 hours: number analyzed (Participants) | 1 | 1
  2 hours | 76.63 (0) | 97.44 (0)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 1 | 1
  end of initial bolus of fluid administration (about 3 hours) | 48.02 (0) | 32.93 (0)
  12 hours: number analyzed (Participants) | 1 | 0
  12 hours | 171.29 (0) |
  24 hours: number analyzed (Participants) | 1 | 1
  24 hours | 97.44 (0) | 215.23 (0)

5. Primary Outcome: Sympatho-adrenal Activation as Assessed by Norepinephrine (NE)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: Data was not collected for one participant at the end of initial bolus of fluid administration (about 3 hours) and 24 hours in the initial resuscitation with balanced crystalloids arm.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours | 3539.75 (3998.06) | 1757.75 (718.80)
  2 hours | 5434.25 (9411.88) | 2877 (2349.24)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 5271 (9131.59) | 2398.33 (1208.69)
  12 hours | 8360.75 (15166.41) | 1643.5 (959.69)
  24 hours: number analyzed (Participants) | 4 | 3
  24 hours | 6579.25 (10412.6) | 1180.33 (899.90)

6. Primary Outcome: Sympatho-adrenal Activation as Assessed by Epinephrine (Epi)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: Data was not collected for one participant at the end of initial bolus of fluid administration (about 3 hours) and 24 hours in the initial resuscitation with balanced crystalloids arm.
  Sample levels were out of range and thus no value could be obtained for one participant at 24 hours in the initial resuscitation with balanced crystalloids arm.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours | 239 (139.90) | 87.25 (42.01)
  2 hours | 198 (145.22) | 132 (34.47)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 226.5 (210.47) | 160.66 (148.39)
  12 hours | 143.75 (113.70) | 138.25 (42.43)
  24 hours: number analyzed (Participants) | 4 | 2
  24 hours | 133 (77.48) | 191 (108.89)

7. Primary Outcome: Inflammation as Assessed by Soluble Receptor for Advanced Glycation Endproduct (sRAGE)
Time Frame: 0, 2, end of initial bolus of fluid administration, 12, and 24 hours
Population: Data was not collected for this outcome measure.
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Inflammation as Assessed by High Mobility Group Protein-1 (HMGB-1)
Time Frame: 0, 2, end of initial bolus of fluid administration, 12, and 24 hours
Population: Data was not collected for this outcome measure.
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Inflammation as Assessed by Interleukin-6 (IL-6)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours | 2455.043 (4421.03) | 782.41 (977.31)
  2 hours | 1911.7 (3571.24) | 189.41 (121.41)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 1911.48 (3587.39) | 109.79 (9.13)
  12 hours | 1076.74 (2062.13) | 60.02 (51.39)
  24 hours: number analyzed (Participants) | 4 | 3
  24 hours | 296.94 (529.58) | 29.27 (20.38)

10. Primary Outcome: Inflammation as Assessed by Interleukin-8 (IL-8)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours) , 12, and 24 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours | 866.78 (1599.38) | 180.46 (184.81)
  2 hours | 695.66 (1276.29) | 93.53 (34.03)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 763.04 (1414.59) | 83.13 (17.28)
  12 hours | 632.78 (1170.42) | 58.84 (11.39)
  24 hours: number analyzed (Participants) | 4 | 3
  24 hours | 158.71 (242.78) | 43.37 (10.80)

11. Primary Outcome: Inflammation as Assessed by Interleukin-10 (IL-10)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: Data was not collected for one participant at the end of initial bolus of fluid administration (about 3 hours) and 24 hours in the initial resuscitation with balanced crystalloids arm.
  Sample levels were out of range and thus no value could be obtained for one participant at 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours in the initial resuscitation with plasma arm.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours | 140.06 (254.38) | 101.88 (183.79)
  2 hours: number analyzed (Participants) | 3 | 4
  2 hours | 216.59 (349.54) | 52.50 (81.70)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 3 | 3
  end of initial bolus of fluid administration (about 3 hours) | 257.11 (422.66) | 84.52 (127.60)
  12 hours: number analyzed (Participants) | 3 | 4
  12 hours | 59.79 (79.01) | 9.20 (3.93)
  24 hours: number analyzed (Participants) | 3 | 3
  24 hours | 23.51 (22.55) | 6.27 (1.20)

12. Primary Outcome: Inflammation as Assessed by Interleukin-1α (IL-1α)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours | 15221.21 (11064.91) | 7759.09 (3512.66)
  2 hours | 11724.06 (8728.74) | 7475.72 (3752.85)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 12305.08 (10084.78) | 7833.37 (4661.07)
  12 hours | 7998.79 (7952.26) | 3770.93 (2453.76)
  24 hours: number analyzed (Participants) | 4 | 3
  24 hours | 5922.11 (6274.24) | 1999.86 (1953.98)

13. Primary Outcome: Inflammation as Assessed by Interleukin-1β (IL-1β)
Time Frame: 0, 2, end of initial bolus of fluid administration (about 3 hours), 12, and 24 hours
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
pg/mL
  0 hours | 17.59 (29.76) | 2.55 (1.64)
  2 hours | 7.21 (10.97) | 1.99 (.98)
  end of initial bolus of fluid administration (about 3 hours): number analyzed (Participants) | 4 | 3
  end of initial bolus of fluid administration (about 3 hours) | 8.31 (13.43) | 2.10 (.81)
  12 hours | 1.95 (1.35) | 1.48 (.44)
  24 hours: number analyzed (Participants) | 4 | 3
  24 hours | 1.56 (.66) | 1.61 (.26)

14. Secondary Outcome: Total Volume of Fluid Required for Resuscitation After the Initial Bolus of Either Plasma or Crystalloids
Description: Data were not collected for 1 participant in the initial resuscitation with plasma arm.
Time Frame: First 24 hours after initiation of fluid resuscitation
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 3 | 4
mL | 967.66 (951.91) | 455 (530.50)

15. Secondary Outcome: Time Until Lactate Normalization
Time Frame: First 24 hours after initiation of fluid resuscitation
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
hours | 15.25 (27.26) | 3.5 (7)

16. Secondary Outcome: Time on Vasopressors
Time Frame: First 30 days after initiation of fluid resuscitation
Population: Data were not collected for 2 participants in the initial resuscitation with plasma arm and 2 participants in the initial resuscitation with balanced crystalloids arm.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 2 | 2
hours | 70.5 (92.63) | 14.5 (10.60)

17. Secondary Outcome: Number of Days on Ventilator Support
Time Frame: First 30 days after initiation of fluid resuscitation
Population: Data were not collected for 1 participant in the initial resuscitation with balanced crystalloids arm.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 3
days | 13.5 (10.37) | 9 (15.58)

18. Secondary Outcome: Number of Intensive Care Unit (ICU)-Free Days
Time Frame: First 30 days after initiation of fluid resuscitation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
days | 9.25 (13.20) | 23.5 (22.53)

19. Secondary Outcome: Number of Hospital Days
Time Frame: From the time of initiation of fluid resuscitation to the time of hospital discharge (up to about 170 days)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
days | 29 (11.16) | 81.5 (86.54)

20. Secondary Outcome: Mortality
Time Frame: First 30 days after initiation of fluid resuscitation
Measure: Count of Participants; unit: Participants
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 4 | 4
Participants | 1 | 1

21. Secondary Outcome: Number of Participants With Acute Lung Injury
Time Frame: First 30 days after initiation of fluid resuscitation
Population: Data was not collected for this outcome measure.
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 0 | 0

22. Secondary Outcome: Number of Participants With Acute Kidney Injury
Time Frame: First 30 days after initiation of fluid resuscitation
Population: Data was not collected for this outcome measure.
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Initial Resuscitation With Plasma | Initial Resuscitation With Balanced Crystalloids
All-Cause Mortality (participants affected / at risk) | 1/4 | 1/4
Serious Adverse Events (participants affected / at risk) | 4/4 | 4/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Initial Resuscitation With Plasma (N=4) | Initial Resuscitation With Balanced Crystalloids (N=4)
Acute Kidney Injury (Renal and urinary disorders) | 0 | 1
Liver failure (Hepatobiliary disorders) | 0 | 1
Clostridium difficile colitis (Gastrointestinal disorders) | 0 | 1
atrial fibrillation requiring multiple cardioversions (Cardiac disorders) | 0 | 1
acute renal failure requiring intermittent hemodialysis (Renal and urinary disorders) | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 1
acute renal failure requiring continuous renal replacement therapy/intermittent hemodialysis (Renal and urinary disorders) | 0 | 1 — (resolved)
acalculous cholecystitis (Hepatobiliary disorders) | 0 | 1
medication induced blindness (Eye disorders) | 0 | 1
Deep vein thrombosis with persistent anemia requiring inferior vena cava filter (Vascular disorders) | 0 | 1
anemia requiring Inferior vena cava filter (Blood and lymphatic system disorders) | 0 | 1
chylothorax (Blood and lymphatic system disorders) | 0 | 1
multiple episodes of severe sepsis secondary to urinary tract infection (Infections and infestations) | 0 | 1
bacteremia (Infections and infestations) | 0 | 1
Gastrointestinal bleed (Gastrointestinal disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Urinary tract infection (Renal and urinary disorders) | 1 | 0
Ascending colon perforation (Gastrointestinal disorders) | 1 | 0
Congestive heart failure exacerbation/flash pulmonary edema (Cardiac disorders) | 1 | 0
Worsening acute kidney injury requiring continuous renal replacement therapy to be restarted (Renal and urinary disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Traumatic brain injury (tracheostomy & percutaneous endoscopic gastrostomy) (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT03366220/Prot_SAP_000.pdf